CLINICAL TRIAL: NCT05020197
Title: Study of the Association Between the Type of Attachment and the Risk of Post-Traumatic Stress Disorder: A Prospective Cohort Study in the Forensic Medicine Department of the Hospices Civils de Lyon
Brief Title: Study of the Association Between the Type of Attachment and the Risk of Post-Traumatic Stress Disorder
Acronym: TRAUMAFFECT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0814
Record Dates: First submitted 2021-07-19; First posted 2021-08-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Attachment; PTSD; risk factor
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: self-questionnaires on attachment and PTSD — The questionnaires (attachement type, PTSD symptoms) are administered face to face at the inclusion visit (at D0-D3). Validated self-questionnaires in French will be sent to the patients, either electronically or by post, according to their choice at D30 and D90. To describe the characteristics of the subjects, socio-demographic data, lifestyle, and medical history will be collected. The questionnaires will be administered three times to study the evolution of the parameters over time.

SUMMARY:
Attachment theory models the emotional bonding that is activated in situations of danger, via mental representations of self and others. Four types of attachment (TA) exist in adults: 3 insecure (Preoccupied, Detached, Fearful) and 1 secure. Attachment type is a major factor in the development of Post-Traumatic Stress Disorder (PTSD), a frequent and disabling mental disorder that occurs after a traumatic event. A meta-analysis based on Anglo-Saxon studies including various populations (general, military or clinical) (n=9268 patients) suggested an association between Fearful BP and high level of PTSD symptoms (r=0.44). Nevertheless, these results did not allow the identification of variations related to the individual risk factors (RDFs) of the subject and his environment, especially in the French socio-cultural context. The investigators propose to study the association between LDs and the risk of PTSD in the days following exposure, their mutual influence in the months following, and their associated factors. Thus, a prospective cohort study among French adult victims of a traumatic event could objectify the link between BP - as close as possible to the event - and the risk of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Having experienced a Potentially Traumatic Event within 3 days and according to DSM5 criterion A: Exposure to actual or potential death, serious injury, or sexual violence in one (or more) of the following ways: Directly experiencing the traumatic event, witnessing the event in person by others, learning that the traumatic event (violent or accidental) was experienced by a close family member or friend, experiencing repeated or extreme exposure to the harrowing details of the traumatic event (e.g., first responders or police officers) (exposure through electronic media, television, films, or photographs, if the exposure is work-related)
* Good understanding of oral and written French
* Having given written consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Psychiatric pathology with current clinical instability (agitation, maladaptive consciousness...) or patient unable to understand questionnaires
* Vulnerable adult (curatorship, guardianship)
* Non French resident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Having experienced a Potentially Traumatic Event within 3 days and according to DSM5 criterion A: Exposure to actual or potential death, serious injury, or sexual violence in one (or more) of the following ways: Directly experiencing the traumatic event, witnessing the event in person by others, learning that the traumatic event (violent or accidental) was experienced by a close family member or friend, experiencing repeated or extreme exposure to the harrowing details of the traumatic event (e.g., first responders or police officers) (exposure through electronic media, television, films, or photographs, if the exposure is work-related)
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Experiences in Close Relationships-Revised (ECR-R) attachment questionnaire | Day 30
  Type of attachment Disorder will be measured at inclusion by the ECR-R attachment questionnaire. Each item is rated on a 7-point scale where 1 = strongly disagree and 7 = strongly agree.
Questionnaire Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Day 30
  Risk of developing Post Traumatic Stress Disorder. Items are rated on a 5 point scale. The maximum score is 80.
Correlation between Questionnaire PCL-5 AND ECR-R attachment questionnaire | Day 30
  Correlation of outcome 1 and outcome 2

SECONDARY OUTCOMES:
Questionnaire Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Day 90
  Risk of Post-Traumatic Stress Disorder at 90 days. Items are rated on a 5 point scale. The maximum score is 80.
Questionnaire Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Day 90
  Type of attachment. Items are rated on a 5 point scale. The maximum score is 80.
Correlation between PCL-5 questionnaire.And PCL-5 questionnaire.at D90 | Day 90
  Correlation between the type of attachment and the risk of Post-Traumatic Stress Disorder
Relationship Scales Questionnaire (RSQ) | Day 3
  30-item self-questionnaire that categorizes participants into four categories of attachment (secure or autonomous, avoiding or detached, preoccupied or ambivalent, fearful or disorganized)
Relationship Scales Questionnaire (RSQ) | Day 30
  30-item self-questionnaire that categorizes participants into four categories of attachment (secure or autonomous, avoiding or detached, preoccupied or ambivalent, fearful or disorganized)
Relationship Scales Questionnaire (RSQ) | Day 90
  Measure of Psychometric performance; 30-item self-questionnaire that categorizes participants into four categories of attachment (secure or autonomous, avoiding or detached, preoccupied or ambivalent, fearful or disorganized)
Experiences in Close Relationships-Revised (ECR-R) attachment questionnaire | Day 3
  Attachment Type. Each item is rated on a 7-point scale where 1 = strongly disagree and 7 = strongly agree
Experiences in Close Relationships-Revised (ECR-R) attachment questionnaire | Day 30
  Attachment Type. Each item is rated on a 7-point scale where 1 = strongly disagree and 7 = strongly agree
Experiences in Close Relationships-Revised (ECR-R) attachment questionnaire | Day 90
  Attachment Type. Each item is rated on a 7-point scale where 1 = strongly disagree and 7 = strongly agree
Questionnaire Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Day 90
  Risk of Post Traumatic Stress Disorder (D90). Items are rated on a 5 point scale. The maximum score is 80.
Impact of Event Scale Revised | Day 3
  The IES-R consists of a list of 22 symptoms of PTSD. The person indicates the intensity with which each symptom has manifested itself over the past 7 days, by self-reporting their response on a 5-point Lykert-type scale, ranging from 0 ("Not at all") to 4 ( "Extremely"). The total IES-R score is calculated by adding the values obtained for the 22 items (scores 0-88).
Relationship Scales Questionnaire (RSQ) | Day 90
  30-item self-questionnaire that categorizes participants into four categories of attachment (secure or autonomous, avoiding or detached, preoccupied or ambivalent, fearful or disorganized)

CONTACTS AND LOCATIONS:
Overall Officials: Ludivine NOHALES, MD, Principal Investigator — Service de médecine et santé au travail des HCL
Locations (1):
- Service de médecine et santé au travail des HCL, Lyon, France